CLINICAL TRIAL: NCT06221033
Title: Manual Hyperinflation Versus Diaphragmatic Proprioceptive Neuromuscular Facilitation on Pulmonary Functions in Mechanically Ventilated Patients
Brief Title: Comparing the Effects of Manual Hyperinflation and Diaphragmatic Proprioceptive Neuromuscular Facilitation on Pulmonary Functions in Patients on Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: omar hasham mohamed (Other)
Responsible Party: Sponsor-Investigator, omar hasham mohamed, physiotherapist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004933
Record Dates: First submitted 2024-01-01; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: COPD Exacerbation Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- manual hyperinflation group (Experimental): this group will receive manual hyper inflation technique as a treatment modality
  Interventions: Device: manual hyperinflation
- diaphragmatic proprioceptive neuromuscular facilitation group (Experimental): this group will receive diaphragmatic proprioceptive neuromuscular facilitation technique
  Interventions: Other: Diaphragmatic proprioceptive neuromuscular facilitation technique
- control group (Other): this group will receive the traditional physiotherapy techniques ( percussion , shaking , breathing ex )
  Interventions: Other: traditional physiotherapy

INTERVENTIONS:
Device: manual hyperinflation — Each participant will assume a relaxed comfortable in supine position. Bag valve resuscitation circuit locked at pressure 35 cm H20 will be used. Six sets of six MHI breaths will be applied. MHI breaths had a slow inspiration for three seconds duration, a three second end inspiratory pause (hold) then an uninterrupted expiration as a quick release
  Arms: manual hyperinflation group
Other: Diaphragmatic proprioceptive neuromuscular facilitation technique — Rhythmic initiation technique that is derived from the PNF concept will be initiated by four 20-second manual diaphragm stimulations. After every stimulation the patient rested for one minute. Therapist's hands will be placed below the rib cage, just below the costal arches and will support patient's exhalation phase by slight lengthening his diaphragm simultaneously in posterior-superior direction using a verbal cue "exhale". At the same time, the patient will verbally be encouraged to take a deep breath
  Arms: diaphragmatic proprioceptive neuromuscular facilitation group
Other: traditional physiotherapy — This group will receive the traditional medical treatment and chest physiotherapy only.
  Arms: control group

SUMMARY:
the goal of this clinical trial is to compare between to important physiotherapy modalities applied on mechanically ventilated COPD patients the the main question the study aim to answer is which one of the two modalities has the better effect on mechanically ventilated patients with COPD

patients will get manual hyperinflation technique and PNF technique \

researchers will compare MHI with PNF and will take a control group also

DETAILED DESCRIPTION:
In this study, the effects of diaphragmatic proprioceptive neuromuscular facilitation and manual hyperinflation on pulmonary functions in patients on mechanical ventilation will be compared.

The following headings will be used to present the study's subject and methods: patients, tools, study protocols, and statistical techniques.

I. Patients

The trial will involve sixty male patients with AECOPD who are on mechanical ventilation. They will be chosen from the Gamal Abdel Nasser Hospital's intensive care unit at the Health Insurance Organization in Alexandria, Egypt. They will be between the ages of fifty and sixty. Three equal groups will be randomly assigned to the study's patients.

Study Group A (20 patients) will undergo chest physiotherapy and conventional medical treatment in addition to manual hyperinflation technique.

Calculating the sample size:

Using G*Power (version 3.1.9.2; Franz Faul, University at Kiel, Germany), the number of patients was determined. This study employed the t-test. Type II error was at 80% power, and type I error was 95% (alpha level: 0.05). The primary dependent variable, arterial blood gases, had an impact size of (Cohen's d) of 0.8. This figure was computed using data from the pilot trial on patients with AECOPD who were on mechanical ventilation. For the purposes of this investigation, sixty patients was the minimum.

Pre-post measures and a single-blinded, randomized controlled trial comprised the study's design. The study will be carried out in the Gamal Abdel Nasser Hospital's intensive care unit at the Health Insurance Organization in Alexandria, Egypt.

Acute exacerbation of chronic obstructive pulmonary disease (AECOPD)

An event in the natural course of the disease known as an exacerbation of COPD is defined as a shift in the patient's baseline dyspnea, cough, and/or sputum that goes beyond daily fluctuation and necessitates a change in treatment.

Tests for pulmonary function (PEFs) A rapid, easy, non-invasive test that measures lung volume, capacity, flow rates, and gas exchange to demonstrate how effectively the lungs are functioning. Consequently, it offers the necessary information that your healthcare professional would need to diagnose and determine the course of treatment for specific lung problems.

manual hyperinflation A high tidal volume can be achieved by manual hyperinflation up to a peak pressure of 40 cmH2O. It begins with a sluggish inspiration, then moves into an inspiratory hold for two or three seconds before rapidly expiring (much like forced expiration). Using a manual hyperinflation bag with a positive end-expiratory pressure (PEEP) valve is one method that helps minimize derecruitment and atelectrauma by maintaining PEEP. Proprioceptive feedback from the bag to the operator is the benefit of manual hyperinflation over ventilator hyperinflation, whereas the safety of PEEP maintenance and the technique's uniformity and reproducibility are the benefits of ventilator hyperinflation. The manual hyperinflation technique is thought to be easier to utilize in awake patients than the ventilator hyperinflation maneuver.

Enhancing mobility of the chest wall can be accomplished by the facilitator technique known as proprioceptive neuromuscular facilitation. The most effective proprioceptive facilitator technique for returning to a normal breathing pattern is intercostal stretch. Other techniques include abdominal cocontraction, moderate manual pressure, perioral pressure, anterior stretch lift to the posterior basal area, and vertebral pressure to the upper and lower thoracic spines. PNF improves muscle strength, endurance, and mobility while facilitating control, stability, and coordinated movement, which sets the groundwork for function restoration.

Pre-post measures and a single-blinded, randomized controlled trial comprised the study's design. The study will be carried out in the Gamal Abdel Nasser Hospital's intensive care unit at the Health Insurance Organization in Alexandria, Egypt.

Ethical considerations:

Each patient and his family will be asked to sign a consent form before the current study begins, indicating their agreement to be part in it. Every patient and his family members will get a thorough explanation of how the assessment and treatment devices work. Each patient and his family will also receive an explanation of the rationale behind the examination and treatment methods

.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included in the study if they have the following criteria:

  1. Sixty male mechanically ventilated patients. They will be ventilated on pressure support (PS) mode of MV with this setting (Positive end-expiratory pressure [PEEP]) less than 8 cm H2O, FiO2 0.4 or less, SpO2 higher than 90) due to AECOPD.
  2. Their Glasgow Coma Scale score will be ranged from 13 to 15.
  3. Their age between 50 and 60 years old.
  4. Their BMI will be ranged from 25 to 34.9 kg/m2.
  5. Moderate (GOLD 2) and severe (GOLD 3) stages of COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) grading system for the severity of COPD.

Exclusion Criteria:

* The patients will be excluded from this study if they have one of the following criteria:

Fever above 38.3 °C. Unstable hemodynamics. Thoracic or abdominal surgery that preclude the use of PNF exercises. Chest trauma such as rib fracture, flail chest and thoracic vertebra fracture or chest burns.

Peripheral and central nervous system diseases. Active lung infection like tuberculosis. Active bleeding as alveolar hemorrhage, hemoptysis. Spinal cord injuries involved the phrenic nerve. Severe cardiac complications due to COPD.

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Blood gases analysis | immediately after the intervention
  Each patient will be informed about the purpose of the test and how it will be done with keeping the explanation brief and in simple terms.
  Each patient will be informed to assume a relaxed comfortable position with loose clothes.
  Arterial blood samples will be taken via arterial line which is accessible and less painful.
  The collected arterial blood sample will be sent for laboratory investigation according to ICU department laboratory communication protocol of Gamal Abdel Nasser Hospital.
  The test will be conducted for all patients pre and post the treatment program duration.
C- reactive protein analysis | immediately after the intervention
  Each patient will be informed about the purpose of the test and how it will be done with keeping the explanation brief and in simple terms.
  Each patient will be instructed to assume a relaxed comfortable position with loose clothes.
  Initial step, phlebotomist will secure a snug rubber band around patient's upper arm, and the patient will be asked to pump his fist several times.
  Then phlebotomist will palpate the vein, and will cleanse with an alcohol prep pad. Then practitioner will introduce a needle into the vein, and will draw a vial of blood.
  After that the practitioner will remove the band, then remove the needle and apply pressure to venipuncture site up to one minute.
  A bandage will be applied over the site. The test will be conducted for all patients pre and post the treatment program duration.
  Normal finding for C-reactive protein (CRP) is < 1.0 mg/dL or <10.0 mg/L (SI units) (< 3 mg/L for high-sensitivity CRP [hs-CRP]),
Assessment of weaning parameters | during the assessment time
  The weaning process will be indicated according to the following criteria; Adequate oxygenation" PaO2/FIO2 ratio ≥ 200, FIO2≤ 0.40, PaO2 ≥ 60, PaCO2 and PEEP ≤ 5 cmH2O", PH ≥ 7.30, Respiratory rate ≤ 45 bpm, Heart rate ≤ 140 bpm, RSBI ≤ 8 breaths/min/ml/kg body weight, Hemodynamic stability" no or minimal vasopressors or inotropes", Appropriate level of conscious, No continuous sedation infusion nor neuromuscular blocking agents, Afebrile, Adequate hemoglobin ≥8 g/dl and/or no evidence of hemorrhage
Oxygenation Index | immediately after the intervention
  Oxygenation index is the better indicator for defining of lung injury compared to the PaO2/FiO2 ratio as it includes mean airway pressure (MAP), also it is an important determinant of oxygenation of acute respiratory failure, which evaluated according the following equation (PaO2/ FiO2) <300 mmHg with or without elevated arterial carbon dioxide tension (PaCO2) (Liu et al., 2015). OI is a commonly used to assess the severity of hypoxic respiratory failure (HRF) and persistent pulmonary hypertension OI = mean airway pressure MAP (in cmH2O) × FiO2 × 100 ÷ PaO2 . Where FiO2: Fraction of inspired oxygen in percent. MAP: Mean airway pressure in mmHg. FiO2: Fraction of inspired oxygen. PaO2: Partial pressure of oxygen in arterial blood in mmHg. The oxygenation index will be recorded for all patients pre and post the treatment program duration.
Assessment of chest expansion | immediately after the intervention
  Each patient will be informed about the purpose of the test and how it will be done with keeping the explanation brief and in simple terms.
  Each patient will assume a comfortable half lying suping position. Marking will be done at 3 levels; axillary, nipple and xiphisterna. Patient will be asked to first take some normal breaths as a breath control technique for relaxation. Then will be asked to exhale completely and then inhale maximally as much as he can and hold breath for a second.
  The difference between maximum exhalation and inhalation will be recorded during holding breath using a measuring tape at all three-level mentioned above. This procedure will be repeated three times and then the best value will be recorded The chest expansion will be measured for all patients pre and post the treatment program duration

SECONDARY OUTCOMES:
Weaning success rate: | immediately after the intervention
  Weaning success defined as spontaneous breathing without mechanical support for at least 48 hours. Weaning success rate, a proportion of successfully weaned patients to total number of patients receiving a treatment program, was recorded for three study groups post the treatment program duration

CONTACTS AND LOCATIONS:
Locations (1):
- Gamal Abdelnasser Hospital, Alexandria, Alexandria Governorate, Egypt